CLINICAL TRIAL: NCT06086392
Title: Effect of Perineural Dexamethasone on the Duration of Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery
Brief Title: Perineural Dexamethasone in Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-01

CONDITIONS: Wrist Disease; Hand Injuries; Wrist Injuries; Hand Disease; Hand Injuries and Disorders
MeSH Terms: conditions — Hand Injuries; Wrist Injuries; Disease | interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Active Comparator): 0.2% ropivacaine for supraclavicular brachial plexus block
  Interventions: Drug: Placebo
- 0.1mg/kg Dexamethasone (Active Comparator): 0,1mg/kg dexamethasone added to 0.2% ropivacaine for supraclavicular brachial plexus block
  Interventions: Drug: 0.1mg/kg Dexamethasone
- 0,05mg/kg dexamethasone (Active Comparator): 0,05mg/kg dexamethasone added to 0.2% ropivacaine for supraclavicular brachial plexus block
  Interventions: Drug: 0.05mg/kg Dexamethasone

INTERVENTIONS:
Drug: Placebo — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the supraclavicular brachial plexus block
  Other Names: 0.9% sodium chloride
  Arms: Placebo
Drug: 0.1mg/kg Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the supraclavicular brachial plexus block
  Other Names: large dose dexamethasone
  Arms: 0.1mg/kg Dexamethasone
Drug: 0.05mg/kg Dexamethasone — administration of 0.5ml/kg of 0,2% ropivacaine with 0.05mg/kg Dexamethasone for the supraclavicular brachial plexus block
  Other Names: small dose dexamethasone
  Arms: 0,05mg/kg dexamethasone

SUMMARY:
Effect of Perineural Dexamethasone on the Duration of Supraclavicular Brachial Plexus Block for Anesthesia After Pediatric Hand/Wrist Surgery

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineurial Dexamethasone on the duration of supraclavicular brachial plexus block for analgesia after pediatric ankle surgery.

After hand and wrist surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare different doses of perineural Dexamethasone. Groups 2 and 3 have dexamethasone doses of 0.1mg/kg and 0.05mg/kg added to local anesthetic.

The investigator's goal is to find a dexamethasone dose that is as low as possible but simultaneously covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for hand/wrist surgery
* body weight > 5kg

Exclusion Criteria:

* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid Consumption | 48 hours
  Total opiate consumption after surgery
Pain score | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  children <3years old FLACC score (Face, Legs, Activity, Cry, Consolability) children >3years old NRS (Numerical Rating Scale)
Blood glucose | 24 and 48 hours after surgery
  Blood glucose every 24 hour during hospitalization
NLR | 24 and 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 24 and 48 hours after surgery
  Platelet-to-lymphocyte ratio
Mobilisation | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  Finger movement every 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Romanowski, Prof.dr hab., Study Director — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Skórzewo, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No